CLINICAL TRIAL: NCT00575796
Title: Weekly Vinblastine for Chemotherapy Naive Children With Progressive Low Grade Glioma (PLGGs)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Pediatric Oncology Group of Ontario (Other); Brain Tumour Program (Other)
Responsible Party: Principal Investigator, Ute Bartels, Staff Physician, Neuro-Oncology, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000011227
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Glioma
Keywords: pediatrics; Low Grade Glioma; Vinblastine
MeSH Terms: conditions — Glioma | interventions — Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Children will be treated with Vinblastine Sulphate chemotherapy via intravenous administration once a week over a period of 26 weeks. MRI disease evaluation should be performed at weeks 12 and 26 (+/- 1 week). If response on MRI at week 26 > stable (i.e. stable disease, objective or partial or complete response compared to the baseline MRI exam), continue weekly Vinblastine to the total duration of treatment (i.e. 70 weeks).
  All children will be followed until they demonstrate clear signs tumour progression.
  Interventions: Drug: Vinblastine Sulphate

INTERVENTIONS:
Drug: Vinblastine Sulphate — Vinblastine dose: 6 mg/m2 (10 mg maximum dose) route intravenous administration once a week.

SUMMARY:
The overall objective of this study is to determine the efficacy of weekly Vinblastine in chemotherapy naïve patients with progressive or incompletely resected paediatric low grade glioma, to generate estimates of the response rate, progression-free survival, toxicity and quality of daily living among the population treated and determine biologic factors which will enable us to predict tumour behaviour.

DETAILED DESCRIPTION:
Unresectable low grade glioma (LGG) of childhood increasingly appears as a chronic condition for which multiple treatments may be required. While several studies have shown evidence of short term tumour control with chemotherapy, the progression-free survival at 5 years is unsatisfactory. In addition, several regimens currently used for this condition are associated with significant risks of side effect and long term toxicity.

We have piloted in a single arm study the feasibility and efficacy of Vinblastine for children with recurrent and refractory low grade glioma, who have failed at least one line of treatment (chemotherapy and/or irradiation). Preliminary results show promising activity with minimal toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have been < 18 years of age when originally diagnosed.
2. Histologic Diagnosis: Patients must have histologic verification of LGG at original diagnosis. Exceptions are optic pathway gliomas in children with neurofibromatosis or children with large hypothalamic tumours for which a diagnostic biopsy does not seem necessary. Patients with disseminated low grade glioma are eligible.

   1. Astrocytoma Variants: fibrillary, protoplasmic, gemistocytic, mixed
   2. Pilocytic Astrocytoma
   3. Pleomorphic Xanthoastrocytoma
   4. Infantile desmoplastic astrocytoma
   5. Ganglioglioma
   6. Oligodendroglioma
   7. Mixed glioma (including oligo-astrocytoma)
   8. Pilomyxoid astrocytoma
3. Performance Level :Patients must have an ECOG performance status of 0, 1 or 2 or a Lansky/Karnofsky score > 50
4. Life expectancy: Patients must have a life expectancy of * 2 months.
5. Prior Therapy: Patients are eligible at the time of diagnosis or first progression following treatment with surgery only.
6. Measurable Disease: Patients must have measurable disease, documented by radiographic criteria.
7. Concomitant Medications

   1. Steroids: Steroids may be used at the time of inclusion to control progressive symptoms.
   2. Anti-epileptic medications are permitted - levetiracetam (Keppra) or clobazam (Frisium) being the preferred anti-epileptic medications for chronic use reserving phenytoin and lorazepam for acute seizure control.
8. Organ Function Requirements: All patients must have adequate organ and bone marrow function within 7 days of starting chemotherapy (ANC * 1.0 x 109/L /, and platelet count * 100 x 109/L (transfusion independent).
9. Regulatory: All patients and/or their parents or legal guardians must sign a written informed consent and all institutional requirements for human studies must be met. This study is open to all participants regardless of gender or ethnicity.

Exclusion Criteria:

Inclusion criteria are restrictive. Patient must meet all inclusion criteria.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
The response rate to weekly vinblastine | 70 Weeks

SECONDARY OUTCOMES:
The progression-free survival with Vinblastine | At one year, two years and three years
The quality of daily life during treatment | 26 Weeks
The correlation of biological features of LGG with tumour behaviour | 5 years
To determine the role of telomere maintenance in the prognosis and evolution of PLGG | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ute Bartels, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada; Bruce Crooks, MD, Study Chair — IWK Health Centre
Locations (17):
- Canada (17):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Hospital Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Sainte-Foy, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Center, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Lassaletta A, Scheinemann K, Zelcer SM, Hukin J, Wilson BA, Jabado N, Carret AS, Lafay-Cousin L, Larouche V, Hawkins CE, Pond GR, Poskitt K, Keene D, Johnston DL, Eisenstat DD, Krishnatry R, Mistry M, Arnoldo A, Ramaswamy V, Huang A, Bartels U, Tabori U, Bouffet E. Phase II Weekly Vinblastine for Chemotherapy-Naive Children With Progressive Low-Grade Glioma: A Canadian Pediatric Brain Tumor Consortium Study. J Clin Oncol. 2016 Oct 10;34(29):3537-3543. doi: 10.1200/JCO.2016.68.1585. PMID 27573663